CLINICAL TRIAL: NCT03926871
Title: Ergonomics Training Program to Novice and Experienced Workers in Poultry Processing Industry: A Quasi-experimental Study
Brief Title: Ergonomics Training Program to Industrial Workers
Acronym: Ergonomics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosimeire Simprini Padula (Other)
Responsible Party: Sponsor-Investigator, Rosimeire Simprini Padula, Adjunt professor, Universidade Cidade de Sao Paulo
Organization: Universidade Cidade de Sao Paulo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 734.500
Record Dates: First submitted 2019-04-16; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Occupational Exposure

STUDY DESIGN:
Intervention Model Description: Two independents groups (Novice and Experienced). Both groups received ergonomics training in workplace.
Who Masked: Outcomes Assessor
Masking Description: The evaluators performed the biomechanical exposure analysis without knowing that the workers were from the novice and experienced group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novices (Experimental): They received ergonomic training after 1-2 days of hiring to do the work in the cutting room, and packaging sectors. They did not have experience in the refrigerator or butchers, so they had the minimum of information about tasks and risks.
  Interventions: Other: Ergonomic Training
- Experienced (Experimental): They received the same ergonomic training as the newbies, and should have been hired for more than 6 months in the company. In this period they had already acquired patterns of movement and self-protection to accomplish the tasks.
  Interventions: Other: Ergonomic Training

INTERVENTIONS:
Other: Ergonomic Training — The ergonomic training consisted of an educational program in Ergonomics with a duration of 60 (sixty) minutes divided into a theoretical exposition and videos of the occupational tasks performed by the workers themselves. Theoretical lecture covered topics such as ergonomics, human anatomy, worker health, prevention measures to minimize the risks of musculoskeletal diseases. A better way of performing the work to protect the musculoskeletal system was demonstrated.
  Other Names: Postural and Occupational (tasks) training

SUMMARY:
This quasi-experimental study was performed in poultry processing industry. The study aimed to evaluate the benefits of ergonomic training for novice and experienced workers. Sociodemographic and occupational questionnaires were evaluated, musculoskeletal complaints and pain intensity, perceived occupational effort, biomechanical exposure and perception in adopting the training. Complaints in the cervical, wrist and lumbar region were reduced with training, but the intensity of pain was only reduced in the wrist region. There was a reduction in the occupational biomechanical exposure from pre-training, to the post-immediate, and from pre-training to after 2 months for both beginners and experienced. The group of novice workers differed from those with the highest biomechanical exposure reduction in the cutting room tasks. All workers were benefited by ergonomic training in the short and medium term.

DETAILED DESCRIPTION:
The research was submitted to the Local Research Ethics Committee and approved by the number 734.500.

Were included 51 employees from the packing and cutting room sectors. The workers were allocated to Novato and Experienced workers groups. The inclusion criteria for the Novato workers group were to be newly hired (1 to 2 days in the company) and not have previous experience in a poultry processing industry, or butcher's shop. It is to ensure that they did not have prior knowledge of the activity. In the case of the group of experienced workers.

The exclusion criteria were they worked on the task for more than six months and not be absent during the study period (scheduled vacations). Workers who had already received ergonomic training, such as general guidelines and postural adjustments, as well as pregnant women and people with disabilities were excluded.

Outcomes measure

1. Musculoskeletal Complains and Pain Intensity The Nordic Musculoskeletal Questionnaire was used to investigate the presence of musculoskeletal symptoms in the last month, using dichotomous responses (yes or no) The visual analogue pain scale evaluated the intensity of symptoms indicating "absence of pain" (0) on one side and the opposite side "unbearable pain" (10 cm) (Carlsson 1982). The QNSO and pain scale were applied in both groups at the baseline, and after 2 months of the ergonomic training program.
2. Biomechanical Exposure Analysis The analysis of occupational biomechanical exposure occurred through a Poultry processing Check list (PPChecklist) created for the study. The PPChecklist evaluation criteria were based on observational methods for biomechanical exposure analysis, such as the Rapid Upper Limb Assessment (RULA) and Strain Index and the Checklist for Musculoskeletal Risk Assessment (RARME).

   The analyzes of the video tasks of each worker for the application of the PPChecklist was performed by two independent evaluators (MSD and DPV) with experience in Worker's Health and Ergonomics. The results obtained with the analysis of the biomechanical exposure of each segment (cervical, shoulder, forearm, wrist, hand and spine) were added to obtain a general task risk score for each worker with a variation of the score between 0 -19 points. The higher the score, the greater the biomechanical exposure of the workers.
3. Perceived effort and Training Perception The effort perceived by workers in pre-training was evaluated by Borg scale ranges from zero (rest / effortless perceived) to ten (very, very heavy / too much, too much effort).

To evaluate the self-perception of the ease / difficulty of following the training guidelines was created a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

To Novato workers

* 1 to 2 days in the company
* Not have previous experience in a frigorifico, or butcher's shop
* Not have prior knowledge of the activity. To experienced workers
* Work on the task for more than six months
* Be present in company during the study period

Exclusion Criteria:

For all workers

* Had already received ergonomic training (general guidelines and postural adjustments)
* Pregnant women
* People with disabilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2014-12-17 (Actual); Study Completion 2015-02-20 (Actual)

PRIMARY OUTCOMES:
Change from Musculoskeletal Complains at 2 months | baseline, after two months
  The Nordic Musculoskeletal Questionnaire was used to investigate the presence of musculoskeletal symptoms in the last month with dichotomous responses (yes or no)
Change from Pain Intensity at 2 months | baseline, after two months
  The visual analogue pain scale evaluated the intensity of symptoms indicating "absence of pain" (0) on one side and the opposite side "unbearable pain" (10 cm).
Change from Biomechanical Exposure immediately after the interventional training and after two months | baseline, after 1-2 days, after two months
  Analysis of the biomechanical exposure of each segment (cervical, shoulder, forearm, wrist, hand and spine) by by an observational method developed for the study with score (0-19 points).

IPD SHARING:
Plan to Share IPD: No